CLINICAL TRIAL: NCT04374461
Title: Phase II Study of N-acetylcysteine in Severe or Critically Ill Patients With Refractory COVID-19 Infection
Brief Title: A Study of N-acetylcysteine in Patients With COVID-19 Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-168
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Covid-19
Keywords: N-acetylcysteine; 20-168
MeSH Terms: conditions — COVID-19 | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is a single-institution study that will be open at MSKCC's Manhattan campus. Patients will be enrolled into 2 separate arms. The mechanically ventilated &/or managed in a critical-care arm is closed to accrual as of September 2020.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- mechanically ventilated &/or managed in a critical-care (Experimental): This arm is closed to accrual as of September 2020. Patients in both arms will receive N-acetylcysteine IV 6 g/day in addition to supportive and/or COVID-19 directed treatments at the discretion of the treating physician.
  Patients will receive treatment for a maximum of 3 weeks or until one of the following:
  Arm A:
  * Transfer out of the critical-care unit
  * Extubation
  * Toxicity
  * Death
  Interventions: Drug: N-acetylcysteine; Other: Peripheral Blood
- non-mechanically ventilated, non-critical-care (Experimental): Patients in both arms will receive N-acetylcysteine IV 6 g/day in addition to supportive and/or COVID-19 directed treatments at the discretion of the treating physician.
  Patients will receive treatment for a maximum of 3 weeks or until one of the following:
  Arm B:
  * Discharge from hospital
  * Admission to a critical-care unit
  * Intubation
  * Toxicity
  * Death
  Interventions: Drug: N-acetylcysteine; Other: Peripheral Blood

INTERVENTIONS:
Drug: N-acetylcysteine — Patients in both arms will receive N-acetylcysteine IV 6 g/day in addition to supportive and/or COVID-19 directed treatments at the discretion of the treating physician. Treatment interruptions for up to 48 hours are permissible if there is a clinical indication to hold the study drug. Patients can restart drug if they have been off drug for less than 48 hours. Patients are also eligible to restart N-acetylcysteine treatment on the same treatment arm without reconsent if they are within the 30 day followup period after their prior course of treatment on this protocol.
Other: Peripheral Blood — A total of 16mL of research whole blood will be collected in CPT tubes at baseline, Cycle 2 Day 1 (or as close as feasible, when still coordinating sample collection across patients in a critical-care unit), and at end of study.

SUMMARY:
The study researchers think that a medication called N-acetylcysteine can help fight the COVID-19 virus by boosting a type of cell in your immune system that attacks infections. By helping your immune system fight the virus, the researchers think that the infection will get better, which could allow the patient to be moved out of the critical care unit or go off a ventilator, or prevent them from moving into a critical care unit or going on a ventilator.

The US Food and Drug Administration (FDA) has approved N-acetylcysteine to treat the liver side effects resulting from an overdose of the anti-inflammatory medication Tylenol® (acetaminophen). N-acetylcysteine is also used to loosen the thick mucus in the lungs of people with cystic fibrosis or chronic obstructive pulmonary disease (COPD). This study is the first to test N-acetylcysteine in people with severe COVID-19 infections.

ELIGIBILITY:
Inclusion Criteria:

* Documented COVID-19 infection (either performed on site or documented external report)
* Age ≥ 18

Arm A:

* Admission to an intensive care unit at MSK (M-11) and/or receiving mechanical ventilation
* Absolute lymphocyte count ≤ 1.0/mm3
* As the ALC of patients with lymphoid malignancies is unreliable, they may be enrolled at the discretion of the treating physician after review of their blood work.

Arm B:

* Arm B:Requiring 2L or more of supplemental oxygen by nasal cannula or higher to maintain SpO2 of 95%

Exclusion Criteria:

Arm B:

* requiring mechanical ventilation or admission to an intensive care unit at MSK (M11)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Arm A: number of patients who are successfully extubated and/or transferred out of critical care due to clinical improvement | 1 year
Arm B: number of patients who are discharged from the hospital due to clinical improvement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santosha Vardhana, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm